CLINICAL TRIAL: NCT03621813
Title: Progressive Activity-Based Rehabilitation in Veteran Cancer Survivors With Chronic Pain
Brief Title: Exercise Rehabilitation in Veteran Cancer Survivors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Baltimore VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: E2870-P; HP-00081388 (Other: Baltimore VAMC)
Record Dates: First submitted 2018-08-03; First posted 2018-08-08 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Cancer
Keywords: Neuropathic Pain; Exercise; Lung Cancer
MeSH Terms: conditions — Neoplasms; Neuralgia; Motor Activity; Lung Neoplasms | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Cancer survivors will be enrolled in a 6-week delayed entry control period followed by 6-week exercise rehabilitation program.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Other): Participants maintain their current activity level.
  Interventions: Other: Control
- Exercise Rehabilitation (Active Comparator): Participants will exercise 2x/week at training facilities and at home one day a week.
  Interventions: Behavioral: Exercise Rehabilitation

INTERVENTIONS:
Behavioral: Exercise Rehabilitation — This training is designed to improve fitness, target the major muscle groups for strength, and to improve balance. Aerobic exercise of walking on a treadmill will be performed. Thera-Bands will be used for resistance exercise for the lower and upper body. Balance program includes core exercises (stepping, weight shifts, etc.) and other progressive exercises.
  Arms: Exercise Rehabilitation
Other: Control — Participants are instructed to maintain current activity level and are monitored for changes.
  Arms: Control

SUMMARY:
Exercise rehabilitation has the potential as a non-pharmacological approach to reduce persistent neuropathic pain in Veterans with lung cancer. By examining the effects of exercise training in Veteran cancer survivors with NSCLC, there is the potential to revolutionize care for a: common, debilitating, and inadequately treated symptom in a growing population. This could lead to a larger investigation to fill critical gaps in the literature and at the same time help discover a new model of care for Veterans with chronic pain. The ultimate goal is to reduce this type of pain for the growing population of cancer survivors while simultaneously reducing the need for problematic opioid management.

DETAILED DESCRIPTION:
Persistent or chronic neuropathic pain, either post-thoracotomy persistent pain (PTPP) or chemotherapy-induced peripheral neuropathy (CIPN) occurs in a majority of lung cancer patients. Thus, not only is this neuropathic pain widespread; there is no way to prevent its development, and long-term use of opioids for control of symptoms could result in addiction. Ultimately, PTPP and CIPN can lead to long-term suffering and disability during the post-treatment phase.(NSCLC), which represents about 85% of lung cancer cases.This is the first project of its kind and the potential impact of this research is large, because exercise training will be a prescription and the first approach for which NSCLC survivors can self-manage chronic neuropathic pain. The ultimate goal of the investigators' work is to reduce neuropathic pain for the growing population of cancer survivors while simultaneously reducing the need for problematic pharmacologic management. Therefore, results of this study have potential for high impact on symptom care because it will allow effective neuropathic pain treatment to be in full control of the Veteran, and likely restore function that is lost during the chronic pain experience.

Specific Aims:

1. To determine the feasibility of conducting an exercise rehabilitation intervention in Veterans with NSCLC and PTPP or CIPN.
2. To determine the effects of a VAMHCS-supervised activity rehabilitation program on chronic pain compared to delayed control.
3. To assess changes in fitness, strength, physical function, fatigue, and quality of life (QoL) after activity-based rehabilitation compared to control period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis with lung cancer
* History of treatment with either thoracotomy procedure or neurotoxic chemotherapy or both
* Completion of thoracotomy or chemotherapy > or = 6 months
* Ability to walk on a treadmill
* Karnofsky performance status > 70
* Score > 1 Neuropathic Pain Scale

Exclusion Criteria:

* Presence of metastatic (stage IV)
* Life expectancy < 6 months
* Musculoskeletal or medical conditions which preclude participation in an exercise program

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain Visual Analog Scale Change | Measured at baseline, after 6 weeks control, and after 6 week intervention
  Scale of 0 (no pain) to 100 (worst imaginable pain)

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement System Neuropathic Pain Quality (PROMIS-PQ Neuro) Change | Measured at baseline, after 6 weeks control, and after 6 week intervention
  0-10 numeric rating
Fitness Change | Measured at baseline, after 6 weeks control, and after 6 week intervention
  VO2peak
Strength Change | Measured at baseline, after 6 weeks control, and after 6 week intervention
  knee extensor strength

CONTACTS AND LOCATIONS:
Overall Officials: Alice S. Ryan, PhD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No